CLINICAL TRIAL: NCT01560520
Title: Physical Activity Immediately After Acute Cerebral Ischemia: Too Little or Too Much?
Brief Title: Physical Activity Immediately After Acute Cerebral Ischemia
Status: Completed | Type: Observational
Sponsor: Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Anna Maria Strømmen, clinical assistant, Hillerod Hospital, Denmark
Other Study IDs: 30704
Record Dates: First submitted 2011-11-02; First posted 2012-03-22 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Ischemic Stroke; Physical Activity
Keywords: acute ischemic stroke; accelerometer
MeSH Terms: conditions — Ischemic Stroke; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Interleukin (IL)-6, IL-1beta, Tumor Nekrosis Factor(TNF)-alpha, C-Reactive Proteine (CRP), IL-1ra, IL-10, fasting-insuline, fasting-glucose
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Accelerometer
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — Observation only
  Other Names: actical, Actical

SUMMARY:
Stroke is the leading cause of adult disability in Europe and United States and the second leading cause of death worldwide and affects more than 10,000 Danes each year.

Studies in a late and stationary phase after stroke have shown that physical rehabilitation is of great importance for survival and physical ability of these patients, however many studies show that patients lie or sit next to their bed under hospitalization for more than 88.5 % of the daily hours. Physical activity in stroke patients has never previously been measured immediately after debut of symptoms; furthermore there is no knowledge about the optimal dose of physical rehabilitation for these patients.

Accelerometers, small measuring devices, are a relatively new way to measure physical activity precisely, and hence it is possible to obtain an objective measure of how active stroke patients are in the first week after admission. The accelerometers measure a variable voltage, depending on the range and intensity of movement. They can measure movement dependent of the placement of the accelerometer, for instance over the hip, arm or leg. Studies confirm their reliability, even in patients with abnormal gait, such as stroke patients.

Another approach of studying the effects of physical activity and rehabilitation is through the examination of biomarkers. Studies have shown that biomarkers released during physical activity can inhibit biomarkers released after tissue injury in the brain, as seen after stroke. These brain biomarkers cause further damage and studies show that the higher the levels, the higher the damage. It is therefore obvious to examine whether physical activity rehabilitation can down regulate this destructive process in patients with stroke.

Clarification of physical activity in stroke patients immediately after debut of symptoms and examination of both the biochemical aspects of physical rehabilitation as well as the optimal dose of physical rehabilitation is of great importance for many patients, their relatives as well as of a great socioeconomic importance.

The purpose of the project is to describe the amount and pattern of physical activity in stroke patients in the first week after admission. The investigators hypothesis is that patients are inactive for most of the time during hospitalization, activity being correlated with severity of stroke, but not with age, BMI and sex.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted with acute ischemic stroke
* age > 18 years

Exclusion Criteria:

* symptoms attributable to other diseases than ischemic stroke
* debut of symptoms > 48 h prior to admission
* consent not given < 24 h of admission
* pregnancy or lactation
* isolation
* bloodsampling generally not possible
* allergy due to accelerometer wear
* ulcers or other skin diseases in the area of accelerometer placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke admitted acutely to a hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
activity counts per day | up to 7 days

SECONDARY OUTCOMES:
Inflammation level | up to 7 days
  biomarker concentration
Disability | up to 7 days
  Scandinavian Stroke Scale score (SSS), National Institutes of Health Stroke Scale score (NIHSS), Glasgow Coma Scale score (GCS), Barthels Index-100 (BI), 10 Meters Walking Test (10MWT), modified Rankin Scale (mRS)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Strømmen, MD, Principal Investigator — Neurologic Department
Locations (1):
- Hillerød Hospital, Hillerød, Denmark

REFERENCES:
- [Derived] Strommen AM, Christensen T, Jensen K. Quantitative measurement of physical activity in acute ischemic stroke and transient ischemic attack. Stroke. 2014 Dec;45(12):3649-55. doi: 10.1161/STROKEAHA.114.006496. Epub 2014 Nov 4. PMID 25370584